CLINICAL TRIAL: NCT00608595
Title: Pilot COX-2 Activity in Early Stage Rectal Cancer -Short Term Administration of Celecoxib (SPORE)
Brief Title: Celecoxib in Treating Patients With Early-Stage Rectal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A Bapsi Chakravarthy, MD, Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0174; VU-VICC-GI-0174
Record Dates: First submitted 2008-01-30; First posted 2008-02-06 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; recurrent rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Celecoxib; Gene Expression Profiling; Immunohistochemistry; Mass Spectrometry; Biopsy; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention/Celecoxib (Experimental): Celecoxib
  Interventions: Drug: celecoxib; Genetic: gene expression analysis; Genetic: protein expression analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: mass spectrometry; Procedure: biopsy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: celecoxib — Will be administered orally 400 mg po BID starting 5 days prior to planned surgical resection.
  Other Names: Celebrex
Genetic: gene expression analysis — not noted
Genetic: protein expression analysis — Not noted
Other: immunohistochemistry staining method — not noted
Other: laboratory biomarker analysis — not noted
Other: mass spectrometry
Procedure: biopsy — At the time of preoperative evaluation by surgeon as well as one week after administration of Celecoxib.
Procedure: neoadjuvant therapy — not noted
Procedure: therapeutic conventional surgery — not noted

SUMMARY:
RATIONALE: Studying samples of tissue, blood, and urine from patients with cancer in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how rectal cancer will respond to treatment with celecoxib.

PURPOSE: This clinical trial is studying how well celecoxib works in treating patients with early-stage rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine cyclooxygenase-2 (COX-2) over-expression in tumor specimens from patients with early-stage rectal cancer.
* Determine whether administration of a COX-2 inhibitor, celecoxib, results in changes in tumor (COX-2 overexpressing) levels of eicosanoids but not in levels in the surrounding normal tissue that is expected not to express COX-2.
* Determine whether surrogate markers of eicosanoid metabolism (i.e., serum VEGF levels, tumor prostaglandin E_2 [PGE_2], and the major urinary metabolite of PGE_2 [PGE-M]) in biological specimens from these patients correlate with changes noted in tumor tissue.
* Determine if there is a greater change in protein and gene expression from pretreatment biopsy levels in patient tumor specimens (COX-2 overexpressing) vs specimens of surrounding normal tissue (expected not to be COX-2 overexpressing).

OUTLINE: Patients receive oral celecoxib twice daily on days 1-5. Patients then undergo planned local excision or definitive radical resection on day 6.

Tumor tissue and normal tissue (at least 5 cm away from the tumor) samples are collected pretreatment. Post-treatment tissue samples are collected along with the surgery. Serum and urine samples are obtained at baseline and after administration of celecoxib. Tumor and normal tissue specimens are analyzed by assays measuring markers of cyclooxygenase-2 (COX-2) activity (i.e., COX-2 mRNA and protein, tumor prostaglandin E_2 [PGE_2], and VEGF). Tissue samples are also assessed by cDNA microarray and imaging mass spectrometry to determine overall changes in gene and protein expression from pretreatment levels. Surrogate markers of COX-2 activity in serum (i.e., VEGF) and urine (i.e., urinary metabolite of PGE_2 [PGE-M]) are also assessed and compared with changes noted in tumor tissue. COX-2 protein levels are determined by immunohistochemistry in patients with limited pretreatment tumor tissue specimens.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary adenocarcinoma of the rectum (to be histologically confirmed upon study entry)

  * Tumor must be at or below the peritoneal reflection
  * The distal border of the tumor is within 12 cm of the anal verge on proctoscopic examination
* Clinically resectable disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* WBC ≥ 4,000/mm³
* Platelet count ≥ 150,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other serious medical illness (other than rectal cancer) that would preclude study therapy
* No psychiatric condition that would preclude informed consent
* No history of allergy to celecoxib or any other NSAIDs, including acetylsalicylic acid (i.e., aspirin), ibuprofen, or indomethacin
* No history of allergy to sulfonamides

Exclusion criteria:

Not noted

PRIOR CONCURRENT THERAPY:

* At least 7 days since prior and no concurrent NSAIDs or other cyclooxygenase-2 inhibitors
* No concurrent warfarin, except low-dose warfarin (i.e., 1 mg/day) administered for prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-07; Primary Completion 2004-05 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Event rate of over-expression of cyclooxygenase-2 | Pre and post 7 days administration of study drug
Percent change of eicosanoid level | Pre and post celecoxib treatment ratio of eicosanoid production
Percent change of VEGF and prostaglandin-M levels | Pre and post celecoxib treatment VEGF and PGE-M levels
Change of gene and protein expression pattern from pre- to post-treatment levels | Pre and post celecoxib treatment

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Veterans Administration, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee